CLINICAL TRIAL: NCT02098499
Title: Haldol/Diphenhydramine Versus Metoclopramide/Diphenhydramine for Treatment of Acute Headache in the ED: A RCT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No recruitment occurred and PI retired
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMCP.2012.0008
Record Dates: First submitted 2014-03-17; First posted 2014-03-28 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Migraine Headaches; Nausea; Restlessness
MeSH Terms: conditions — Migraine Disorders; Nausea; Psychomotor Agitation | interventions — Haloperidol; Metoclopramide; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haloperidol and Diphenhydramine (Active Comparator): Haloperidol 5mg IV X1 and Diphenhydramine 25mg IV X1
  Interventions: Drug: Haloperidol; Drug: Diphenhydramine
- Metoclopramide and Diphenhydramine (Active Comparator): Metoclopramide 10mg IV X1 and Diphenhydramine 25mg IV X1
  Interventions: Drug: Metoclopramide 10mg; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Haloperidol — 5mg IV
  Other Names: Haldol
  Arms: Haloperidol and Diphenhydramine
Drug: Metoclopramide 10mg — 10mg IV
  Other Names: Reglan
  Arms: Metoclopramide and Diphenhydramine
Drug: Diphenhydramine — 25mg IV
  Other Names: Benadryl

SUMMARY:
Haloperidol is known to be a safe alternative medication to control difficult pain, and has been shown effective when compared to placebo for controlling headaches. Investigators hypothesized that the combination of haloperidol and diphenhydramine would be a useful medication choice for migraine headache patients in the emergency department in comparison to a common migraine treatment regimen of metoclopramide and diphenhydramine.

DETAILED DESCRIPTION:
Investigators conducted a prospective, double-blind, randomized controlled trial in migraine patients who presented to an academic emergency department between June 2013 and November 2013. Research data was derived from an IRB approved protocol. All subjects met IHS migraine criteria and received a one liter bolus of normal saline plus 25 milligrams (mg) of diphenhydramine. Subjects were subsequently randomized to receive 10 mg metoclopramide or 5 mg haloperidol IV. Pain was self-reported at onset and at 20 minute intervals using a 100mm visual analog scale (VAS). Adequate pain control was considered to be patient satisfaction with symptomatic relief. If adequate pain relief was not obtained after 80 minutes, rescue medication was given at the treating physician's discretion. Adverse reactions were recorded and electrocardiograms (ECGs) were obtained before and after study medication administration. Follow up phone surveys were performed 72 hours after discharge to assess headache recurrence, adverse effects, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Migraine Headache must contain the following:

* At least two: Unilateral, Throbbing, Worsening with activity, Moderate to severe pain
* At least one: Nausea or Vomiting, Photophobia or phonophobia
* Ages 18-50

Exclusion Criteria:

* Hypersensitivity to haloperidol, metoclopramide, and/or diphenydramine
* History of ischemic heart disease or signs or symptoms of ischemic heart disease
* History of stroke or transient ischemic attack (TIA)
* History of peripheral vascular disease
* History of uncontrolled hypertension with presenting diastolic blood pressure > 100
* Use of an ergotamine derivatives, triptan, or dopamine-blocking anti-emetic within the past 24 hrs
* Concurrent administration or within 2 weeks of discontinuing an MAO inhibitor
* Concurrent management of hemiplegic or basilar migraine or known neurologic disorder
* Severe hepatic impairment
* Pregnancy or breastfeeding
* History of cancer (except non-melanoma skin cancer)
* Previous involvement in the study
* Febrile to 100.5 or greater
* Any indication for further diagnostic evaluation of this headache such as a lumbar puncture or CT scan.
* Headache differs from their normal headache

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2015-02-11 (Actual); Study Completion 2015-02-11 (Actual)

PRIMARY OUTCOMES:
Pain scores on the visual analog scale | 20, 40, 60, and 80 min after administration of medications, and then again at the 48-72 hour mark

SECONDARY OUTCOMES:
Nausea and restlessness scores on the visual analog scales | 20, 40, 60, and 80 minutes s/p administration of medications, and again 48-72 hours later

OTHER OUTCOMES:
QT prolongation caused by the administration of Haloperidol | 2 hours after administration of Haldol
  EKGs were performed prior to the administration of study meds and then again at the completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gaffigan, MD, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States